CLINICAL TRIAL: NCT02899000
Title: Efficacy and Safety of Adapalene 0.3%/Benzoyl Peroxide 2.5% Gel Plus Doxycycline in Severe Inflammatory Acne (Non-Nodulocystic) Subjects
Brief Title: A Treatment for Severe Inflammatory Acne Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.SPR.US10355
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Results first posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2016-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Benzoyl Peroxide; Adapalene, Benzoyl Peroxide Drug Combination; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acne treatment (Experimental): Topical adapalene 0.3% / benzoyl peroxide 2.5% emulsion gel (one application daily for 12 weeks)
  Oral doxycycline hyclate, 200 mg per day (two 50-mg tablets twice daily for 12 weeks)
  Interventions: Drug: Adapalene 0.3% / benzoyl peroxide 2.5% emulsion gel; Drug: Oral doxycycline hyclate

INTERVENTIONS:
Drug: Adapalene 0.3% / benzoyl peroxide 2.5% emulsion gel — Topical acne therapy
  Other Names: Epiduo Forte
Drug: Oral doxycycline hyclate — Tetracycline-class oral antibacterial 200 mg daily (2 tablets [50 mg], twice daily)

SUMMARY:
Demonstrate that a daily treatment regimen of adapalene 0.3%/benzoyl peroxide 2.5% gel + oral Doxycycline 200 mg is effective and safe in severe inflammatory acne with 3 or fewer nodules or cysts (non-nodulocystic) during a 12-week treatment period.

DETAILED DESCRIPTION:
This Phase 4, 12-week, single-arm, open-label, multi-center investigational efficacy and safety study was conducted in subjects with severe inflammatory acne. Subjects who met the inclusion criteria and none of the exclusion criteria at the Screening visit returned to the clinic for baseline measures (Week 0) and to start treatment, which continued for up to 12 weeks.

Treatment consisted of 2 investigational study drugs:

* A/BPO 0.3%/2.5% gel applied to dry skin as directed by study staff once daily for 12 weeks, at night after washing.
* Doxycycline hyclate 200 mg: each subject was to take 2 50-mg tablets of doxycycline hyclate in the morning and 2 at night, for a total of 4 tablets (a total of 200 mg) daily for 12 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female subjects, 12 years of age or older at Screening visit.
2. Subjects with a clinical diagnosis of severe inflammatory acne (IGA score of 4).
3. Subjects with 4 or fewer nodules or cysts > 1 cm in diameter on the face.
4. Subjects 18 years of age or older must read and sign the Informed Consent Form, which includes Photography Consent and HIPAA authorization, prior to any participation in the study. Consent will be obtained prior to any study-related procedures. Subjects under the age of 18 years must sign an Assent to Participate Form to participate in the study and must have one parent or guardian read and sign the Informed Consent Form prior to any study-related procedure. (The parent or guardian is not required to attend the following visits unless requested.)

Key Exclusion Criteria:

1. Subjects with nodulocystic or conglobate acne, acne fulminans, or secondary acne (chloracne, drug-induced acne, etc.).
2. Subjects with 5 or more acne nodules or cysts > 1 cm in diameter on the face at Screening and Baseline visits.
3. Female subjects who are pregnant, nursing, or planning a pregnancy during the study.
4. Subjects who have used any systemic therapy directed at improving acne, including antibiotics, within 30 days prior to Baseline visit.
5. Subjects who are at risk in terms of precautions, warnings, and contraindications for the investigational study drugs (see Appendix 14.1 for package inserts for adapalene 0.3%/benzoyl peroxide 2.5% gel and doxycycline hyclate Tablets).
6. Subjects with any other condition or circumstance which, in the Investigator's opinion, may put the subject at risk (e.g., a history of significant renal disease with impairment of renal function), confound the study results, or interfere with the subject's participation in the study.
7. Sponsor and study site staff, relatives of staff members, or other individuals who would have access to the clinical study protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-06-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Galderma Laboratories, LP, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Del Rosso JQ, Stein Gold L, Johnson SM, Rueda MJ, Baldwin H, Lain EL, Landis M, Rendon M, Tanghetti E, Weiss J. Efficacy and Safety of Adapalene 0.3%/Benzoyl Peroxide 2.5% Gel Plus Oral Doxycycline in Subjects With Severe Inflammatory Acne Who Are Candidates for Oral Isotretinoin. J Drugs Dermatol. 2018 Mar 1;17(3):264-273. PMID 29537444

RESULTS

PARTICIPANT FLOW:
Groups:
- Acne Treatment: Topical adapalene 0.3% / benzoyl peroxide 2.5% emulsion gel (one application daily for 12 weeks)
  Oral doxycycline hyclate, 200 mg per day (two 50-mg tablets twice daily for 12 weeks)
  Adapalene 0.3% / benzoyl peroxide 2.5% emulsion gel: Topical acne therapy
  Oral doxycycline hyclate: Tetracycline-class oral antibacterial 200 mg daily (2 tablets [50 mg], twice daily)
Period: Overall Study
Arm/Group | Acne Treatment
Started | 186
Completed | 157
Not Completed | 29

BASELINE CHARACTERISTICS:
Population: Safety Population, defined as all subjects who received at least one dose of a study drug, based on drug accountability data. Safety Population n = 175.
Arm/Group | Acne Treatment
Number analyzed (Participants) | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.6 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33
  Not Hispanic or Latino | 142
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 139
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 175
IGA 4 (Investigator's Global Assessment Score) [Count of Participants; unit: Participants] — Investigator's Global Assessment Severity Scale
  IGA0 Clear------------Clear skin with no inflammatory/non-inflammatory lesions.
  IGA1 Almost Clear - A few scattered comedones and a few small papules.
  IGA2 Mild--------------Easily recognizable; less than half the face is involved. Some comedones and some papules/pustules.
  IGA3 Moderate-------More than half of the face is involved. Many comedones, papules/pustules. One small nodule may be present.
  IGA4 Severe----------Entire face is involved. Covered with comedones, numerous papules/pustules. Few nodules may or may not be present.
  Participants | 175
Total Lesion Count [Mean (Standard Deviation); unit: Lesion Count] | 108.1 (48.43)
Inflammatory Lesion Count [Mean (Standard Deviation); unit: Lesion Count] | 44.1 (21.29)
Non-inflammatory Lesion Count [Mean (Standard Deviation); unit: Lesion Count] | 63.9 (38.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Inflammatory Lesions
Description: Change in Number of Inflammatory Lesions from baseline.
Time Frame: Week 12
Population: Intent-to-Treat (ITT) Population: The ITT Population consisted of the entire population enrolled at Baseline. All efficacy data were analyzed for the ITT Population. Baseline lesion counts missing for one patient.
Measure: Mean (Standard Deviation); unit: Inflammatory lesions
Arm/Group | Acne Treatment
Number analyzed (Participants) | 185
Inflammatory lesions | -30.1 (22.3)

2. Secondary Outcome: Number and Percent of Subjects With IGA Success
Description: IGA Success is defined as an IGA rating of Clear (Grade 0) or Almost Clear (Grade 1)
Time Frame: Weeks 4, 8, and 12
Population: Intent-to-Treat (ITT) Population: The ITT Population consisted of the entire population enrolled at Baseline. All efficacy data were analyzed for the ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Acne Treatment
Number analyzed (Participants) | 186
Participants
  Week 4 | 9
  Week 8 | 44
  Week 12 | 69

3. Secondary Outcome: Percent Change From Baseline in Total Lesion Count
Description: Percent Change From Baseline in Total Lesion Count.
Time Frame: Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change in lesions
Arm/Group | Acne Treatment
Number analyzed (Participants) | 185
percent change in lesions
  Week 4 | -38.9 (28.5)
  Week 8 | -53.9 (30.3)
  Week 12 | -62.6 (31.9)

4. Secondary Outcome: Change From Baseline in Total Lesion Count
Description: Change From Baseline in Total Lesion Count.
Time Frame: Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in lesions
Arm/Group | Acne Treatment
Number analyzed (Participants) | 185
change in lesions
  Week 4 | -43.7 (39.4)
  Week 8 | -59.4 (46.5)
  Week 12 | -69.2 (49.6)

5. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion Count
Description: Percent Change From Baseline in Inflammatory Lesion Count.
Time Frame: Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change in lesions
Arm/Group | Acne Treatment
Number analyzed (Participants) | 185
percent change in lesions
  Week 4 | -38.5 (37.9)
  Week 8 | -55.0 (31.9)
  Week 12 | -66.2 (30.5)

6. Secondary Outcome: Change From Baseline in Inflammatory Lesion Count
Description: Change From Baseline in Inflammatory Lesion Count.
Time Frame: Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in lesions
Arm/Group | Acne Treatment
Number analyzed (Participants) | 185
change in lesions
  Week 4 | -18.9 (19.6)
  Week 8 | -25.9 (22.2)
  Week 12 | -30.1 (22.3)

7. Secondary Outcome: Percent Change From Baseline in Non-Inflammatory Lesion Count
Description: Percent Change From Baseline in Non-Inflammatory Lesion Count.
Time Frame: Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change in lesions
Arm/Group | Acne Treatment
Number analyzed (Participants) | 185
percent change in lesions
  Week 4 | -34.6 (45.6)
  Week 8 | -50.2 (36.9)
  Week 12 | -58.7 (38.8)

8. Secondary Outcome: Change From Baseline in Non-Inflammatory Lesion Count
Description: Change From Baseline in Non-Inflammatory Lesion Count.
Time Frame: Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in lesions
Arm/Group | Acne Treatment
Number analyzed (Participants) | 185
change in lesions
  Week 4 | -24.9 (28.4)
  Week 8 | -33.6 (33.0)
  Week 12 | -39.1 (36.2)

9. Secondary Outcome: Investigator's Evaluation: Number of Subjects Not Considered to be Oral Isotretinoin Candidates
Description: At each visit, subjects were evaluated by the investigator to determine whether (in the opinion of the investigator) they would consider them as candidates for oral isotretinoin therapy.
  The outcome measure reports the number and % of subjects who, in the opinion of the investigator, were not considered to be "a candidate for oral isotretinoin therapy."
Time Frame: Weeks 0, 4, 8, and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Acne Treatment
Number analyzed (Participants) | 186
Participants
  Week 0 | 0
  Week 4 | 78
  Week 8 | 121
  Week 12 | 149

10. Secondary Outcome: Subject Assessment of Acne Improvement
Description: Subject Assessment of Acne Improvement on a 6 point scale (0 = Complete Improvement, 1 = Marked Improvement, 2 = Moderate Improvement, 3 = Minimal Improvement, 4 = No Change, 5 = Worse).
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acne Treatment
Number analyzed (Participants) | 186
score on a scale | 1.3 (0.9)

11. Secondary Outcome: Number and Percent of Adverse Events
Description: Number and percent of subjects with any Treatment-Related Adverse Event
Time Frame: Week 12
Population: The Safety Population consisted of the ITT Population following exclusion of subjects who never took the treatment with certainty, based on drug accountability data. All safety analyses were summarized for the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Acne Treatment
Number analyzed (Participants) | 175
Participants | 27

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: Throughout the course of the study, all AEs were monitored and recorded along with date of onset, severity, relationship to study treatment, and outcome.
Arm/Group | Acne Treatment
All-Cause Mortality (participants affected / at risk) | 0/175
Serious Adverse Events (participants affected / at risk) | 0/175
Other Adverse Events (participants affected / at risk) | 22/175
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acne Treatment (N=175)
Nausea (Gastrointestinal disorders) | 4
Headache (Nervous system disorders) | 7
Erythema (Skin and subcutaneous tissue disorders) | 5
Skin burning sensation (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT02899000/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT02899000/SAP_001.pdf